CLINICAL TRIAL: NCT03316469
Title: Circulating Anti-mullerian Hormone as Predictor of Ovarian Response to Clomiphene Citrate in Women With Polycystic Ovary Syndrome
Brief Title: Anti-Mullerian Hormone as Predictor of Ovarian Responce to Clomiphene Citrate in PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Narges Essam El-din Marrey, Resident of obs & gyn., Ain Shams University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Narges Essam protocol 2017
Record Dates: First submitted 2017-10-10; First posted 2017-10-20 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Anti-mullerian hormone
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Clomiphene

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: CC & ovulation (Experimental): AMH level is measured before Clomiphene citrate 100 mg daily for 5 days & detecting Follicular growth assessment by TVU will be performed at day 12 of the menstrual period. Successful and unsuccessful follicular growth will be compared according to the subjects' respective AMH levels.
  Interventions: Drug: Clomiphene Citrate; Diagnostic Test: Follicular growth
- Group B: CC & no ovulation (Experimental): AMH level is measured before Clomiphene citrate 100 mg daily for 5 days & detecting Follicular growth assessment by TVU will be performed at day 12 of the menstrual period. Successful and unsuccessful follicular growth will be compared according to the subjects' respective AMH levels.
  Interventions: Drug: Clomiphene Citrate; Diagnostic Test: Follicular growth

INTERVENTIONS:
Drug: Clomiphene Citrate — 100 mg daily will be provided to the subjects to be taken for 5 days starting from day 2 of their spontaneous periods
  Other Names: Clomide
Diagnostic Test: Follicular growth — Follicular growth assessment by TVU will be performed at day 12 of the menstrual period.

SUMMARY:
Polycystic ovary syndrome (PCOS) is found in 5% to 6% of women of reproductive age. It affects women's reproductive capability; thus patients have risks of infertility, miscarriage, and complicated pregnancy. A study revealed that the prevalence of oligoovulation or anovulation in patients with PCOS ranged from 65% to 80%. Anti-Mullerian Hormone (AMH) is an important regulator in the ovary that play a rule during development and function. It is suspected to affect clomiphene citrate (cc) resistance. In this study the investigator will assess the accuracy of AMH prediction of response to cc in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with PCOS
* Women 20-35 years old.
* BMI ≤30 kg/m without previous ovulation induction.
* Partners with normal semen parameters Parameter World Health Organization (WHO) 2010 Volume1.5 ml Concentration 15 million/ml Progressive motility 32% Normal forms 4%

Exclusion Criteria:

* Women with evidence of hyper-or hypothyroidism, hyperprolactinemia, Cushing's syndrome, congenital adrenal hyperplasia or androgen-secreting tumors.
* Women with factors of infertility other than PCOS
* Women with incomplete data.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
AMH in prediction of Ovulation in women with PCOS. | 10 days
  AMH level is measured 10 days before expected date of ovulation then correlated to ovulation either successfully or not.

REFERENCES:
- [Background] Azziz R. Controversy in clinical endocrinology: diagnosis of polycystic ovarian syndrome: the Rotterdam criteria are premature. J Clin Endocrinol Metab. 2006 Mar;91(3):781-5. doi: 10.1210/jc.2005-2153. Epub 2006 Jan 17. PMID 16418211
- [Background] Catteau-Jonard S, Pigny P, Reyss AC, Decanter C, Poncelet E, Dewailly D. Changes in serum anti-mullerian hormone level during low-dose recombinant follicular-stimulating hormone therapy for anovulation in polycystic ovary syndrome. J Clin Endocrinol Metab. 2007 Nov;92(11):4138-43. doi: 10.1210/jc.2007-0868. Epub 2007 Aug 14. PMID 17698904
- [Background] Dumesic DA, Lesnick TG, Stassart JP, Ball GD, Wong A, Abbott DH. Intrafollicular antimullerian hormone levels predict follicle responsiveness to follicle-stimulating hormone (FSH) in normoandrogenic ovulatory women undergoing gonadotropin releasing-hormone analog/recombinant human FSH therapy for in vitro fertilization and embryo transfer. Fertil Steril. 2009 Jul;92(1):217-21. doi: 10.1016/j.fertnstert.2008.04.047. PMID 18675414
- [Background] Eijkemans MJ, Imani B, Mulders AG, Habbema JD, Fauser BC. High singleton live birth rate following classical ovulation induction in normogonadotrophic anovulatory infertility (WHO 2). Hum Reprod. 2003 Nov;18(11):2357-62. doi: 10.1093/humrep/deg459. PMID 14585887
- [Background] Hart R, Norman R. Polycystic ovarian syndrome--prognosis and outcomes. Best Pract Res Clin Obstet Gynaecol. 2006 Oct;20(5):751-78. doi: 10.1016/j.bpobgyn.2006.04.006. Epub 2006 Jun 12. PMID 16766228
- [Background] Ghobadi C, Nguyen TH, Lennard MS, Amer S, Rostami-Hodjegan A, Ledger WL. Evaluation of an existing nomogram for predicting the response to clomiphene citrate. Fertil Steril. 2007 Mar;87(3):597-602. doi: 10.1016/j.fertnstert.2006.10.002. Epub 2006 Dec 6. PMID 17156783
- [Background] Imani B, Eijkemans MJ, te Velde ER, Habbema JD, Fauser BC. Predictors of patients remaining anovulatory during clomiphene citrate induction of ovulation in normogonadotropic oligoamenorrheic infertility. J Clin Endocrinol Metab. 1998 Jul;83(7):2361-5. doi: 10.1210/jcem.83.7.4919. PMID 9661609
- [Background] Kurabayashi T, Suzuki M, Fujita K, Murakawa H, Hasegawa I, Tanaka K. Prognostic factors for ovulatory response with clomiphene citrate in polycystic ovary syndrome. Eur J Obstet Gynecol Reprod Biol. 2006 Jun 1;126(2):201-5. doi: 10.1016/j.ejogrb.2005.11.005. Epub 2005 Dec 7. PMID 16337728
- [Background] Laven JS, Mulders AG, Visser JA, Themmen AP, De Jong FH, Fauser BC. Anti-Mullerian hormone serum concentrations in normoovulatory and anovulatory women of reproductive age. J Clin Endocrinol Metab. 2004 Jan;89(1):318-23. doi: 10.1210/jc.2003-030932. PMID 14715867
- [Background] Mashiach R, Amit A, Hasson J, Amzalzg S, Almog B, Ben-Yosef D, Lessing JB, Limor R, Azem F. Follicular fluid levels of anti-Mullerian hormone as a predictor of oocyte maturation, fertilization rate, and embryonic development in patients with polycystic ovary syndrome. Fertil Steril. 2010 May 1;93(7):2299-302. doi: 10.1016/j.fertnstert.2009.01.125. Epub 2009 Mar 3. PMID 19261276
- [Background] Messinis IE. Ovulation induction: a mini review. Hum Reprod. 2005 Oct;20(10):2688-97. doi: 10.1093/humrep/dei128. Epub 2005 Jul 8. PMID 16006478
- [Background] Hintze, J. (2011). PASS 11. NCSS, LLC. Kaysville, Utah, USA.
- [Background] Balen A. Ovulation induction. Obstet Gynaecol Reprod Med. 2004;14:261-268.